CLINICAL TRIAL: NCT03958474
Title: Neurobehavioral Mechanisms of Choice in Opioid Use Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joshua A. Lile, Ph.D. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Joshua A. Lile, Ph.D., Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 47844; R01DA047368 (NIH)
Record Dates: First submitted 2019-05-16; First posted 2019-05-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Oxycodone; Remifentanil

STUDY DESIGN:
Intervention Model Description: Within-subjects design
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active treatment followed by placebo treatment (Experimental): Participants complete a gambling task during oxycodone administration and then complete the same gambling task during placebo administration. Participants with a history of IV opioid use can opt to complete a final remifentanil dose-ranging session.
  Interventions: Drug: Oxycodone; Drug: Remifentanil
- Placebo treatment followed by active treatment (Experimental): Participants complete a gambling task during placebo administration and then complete the same gambling task during oxycodone administration. Participants with a history of IV opioid use can opt to complete a final remifentanil dose-ranging session.
  Interventions: Drug: Oxycodone; Drug: Remifentanil

INTERVENTIONS:
Drug: Oxycodone — Participants receive oxycodone or placebo.
Drug: Remifentanil — Participants with a history of IV opioid use can opt to complete a session in which they receive remifentanil.

SUMMARY:
The objective of this protocol is to use probabilistic reinforcement learning choice tasks and magnetic resonance neuroimaging to demonstrate the impact of problematic opioid use and opioid withdrawal on dynamic decision-making and reveal the neurobehavioral and neurobiological processes underlying abnormal task performance. A second objective is to identify an appropriate dose of intravenous remifentanil for subsequent studies in physically dependent individuals with opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Must meet moderate/severe criteria for moderate/severe opioid use disorder, report recent prescription or illicit opioid use, and be opioid dependent, as evidenced by either a urine sample positive for recent opioid use or being in frank withdrawal during screening.
* Female subjects must be using an effective form of birth control (e.g., birth control pills, surgical sterilization, IUD, cervical cap with a spermicide, or abstinence).
* Able to speak and read English
* Subjects who are interested in completing the remifentanil dose-ranging session must report a history of intravenous opioid use and a baseline O2 saturation of 95% or greater.

Exclusion Criteria:

* History of, or current, clinically significant physical disease (e.g., respiratory disease [asthma, COPD, sleep apnea], impaired cardiovascular functioning, seizure disorder or CNS tumors) or current or past history of psychiatric disorder that would limit compliance in the studies, other than substance use disorder.
* Meet diagnostic criteria for psychoactive substance use disorder for substances other than opioids (OUD subjects only) or nicotine that would require detoxification (i.e., alcohol, benzodiazepines or barbiturates).
* Contraindications for MRI scanning (e.g., pacemaker, metal implants, claustrophobia, or any other implanted medical device).
* Vision or hearing problems that would preclude completion of experimental tasks.
* At risk for respiratory complications and have predictors of difficult bag mask ventilation (e.g., dentures, very full beard), in case emergency respiratory intervention is needed.
* Seeking treatment for SUD.
* Poor venous access (only subjects who will participate in the remifentanil dose-ranging session).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Gambling task | Change in monetary rewards earned on a gambling task as a function of the intervention will be assessed by administering this task once per session across two sessions during a 9-day inpatient enrollment in each subject
  The number of monetary rewards earned on a gambling task, in which two options signaled by distinct cues are presented on a computer screen and choosing either could result in the delivery of money, but the reinforcement probabilities of the options differ, and change during the task.

CONTACTS AND LOCATIONS:
Overall Officials: JOSHUA LILE, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT03958474/ICF_000.pdf